CLINICAL TRIAL: NCT06858449
Title: NeoChemoPRT: A Randomized Study of Resistance Training and Post-Workout Protein to Improve Body Composition During Neoadjuvant Chemotherapy for Breast Cancer
Brief Title: Resistance Training and Post Workout Protein to Improve Body Composition During Neoadjuvant Chemotherapy for Breast Cancer
Acronym: NeoChemoPRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Colin Champ, MD, Principal Investigator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-149-SG
Record Dates: First submitted 2025-02-14; First posted 2025-03-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Cancer; Breast Cancer
Keywords: exercise; resistance training
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Motor Activity | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20 grams of protein (Experimental): Participants will be randomized (like flipping a coin) to a post-workout protein consisting of 20 grams of whey protein. The protein will be 100% cold processed and micro-filtered, non-GMO grass-fed whey protein isolate, soy and gluten free, unflavored, and unsweetened. This will include Irish Dairy, which is whey protein isolate and soy lecithin, and Raw GrassFed Whey, which is whey protein concentrate. Participants will not know which amount of protein they receive.
  Interventions: Dietary Supplement: Whey protein (20 grams)
- 60 grams of protein (Experimental): Participants will be randomized (like flipping a coin) to a post-workout protein consisting of 60 grams of whey protein. The protein will be 100% cold processed and micro-filtered, non-GMO grass-fed whey protein isolate, soy and gluten free, unflavored, and unsweetened. This will include Irish Dairy, which is whey protein isolate and soy lecithin, and Raw GrassFed Whey, which is whey protein concentrate. Participants will not know which amount of protein they receive.
  Interventions: Dietary Supplement: Whey protein (60 grams)

INTERVENTIONS:
Dietary Supplement: Whey protein (20 grams) — 20 grams of whey protein
  Arms: 20 grams of protein
Dietary Supplement: Whey protein (60 grams) — 60 grams of whey protein.
  Arms: 60 grams of protein

SUMMARY:
In this study, the investigators hypothesize that a high dose of post-workout protein nutrition regimen focused on food quality and an observed exercise regimen utilizing high-load resistance training initiated during or after cancer treatment will improve body composition and functional capacity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-89 years
2. Women with a biopsy proven diagnosis of invasive carcinoma of the breast.
3. Women must undergo neoadjuvant chemotherapy for breast cancer treatment prior to surgery
4. Must be able to read and understand English and consent for themselves.

Exclusion Criteria:

1. Inability to get up and down off the ground or squat body weight
2. Inability to safely engage in group exercise sessions as deemed by study PI
3. Severe arthritic, joint, cardiovascular, musculoskeletal, or any other condition deemed by PI to be unsafe to engage in resistance training
4. Lactose intolerance
5. Cow's milk or whey protein allergy
6. Pregnant women
7. Males

Ages: 20 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Changes in muscle mass and fat mass (pounds) at completion of chemotherapy | Baseline and at program completion (within 4 weeks of exercise completion).

SECONDARY OUTCOMES:
Response to Chemotherapy Assed Via the Guidelines or the Response evaluation criteria in solid tumors (RECIST) | Chemotherapy response assessment is at program completion (within 4 weeks of exercise completion)
  Response to chemotherapy will be assessed via the guidelines or the Response evaluation criteria in solid tumors (RECIST) criteria version 1.1 before and after chemotherapy with radiographic interpretation on either MRI of the breast or, if unable to get an MRI, PET/CT scan.
Changes in EuroQol-5 Dimensions (EQ-5D) at completion of chemotherapy assessment | Baseline assessment (prior to program) and at exercise program completion (at 24 weeks).
  EuroQol-5 Dimensions-5 Levels total score for the 5 questions ranges from 5 (no problems on any dimension) to 25 (extreme problems on all dimensions). This is calculated by assigning scores of 1 (minimum), 2, 3, 4, and 5 (maximum), to the response categories of "no problems", "slight problems", "moderate problems", "severe problems", and "extreme problems"/"unable to", respectively. Higher scores mean worse outcomes.
Changes in Patient Health Questionnaire-9 (PHQ9) depression score at completion of chemotherapy assessment | Baseline assessment (prior to program) and at exercise program completion (at 24 weeks).
  Patient Health Questionnaire-9 total score for the 9 questions ranges from 0 (no depression) to 27 (highest level of depression). This is calculated by assigning scores of 0 (minimum), 1, 2, and 3 (maximum), to the response categories of "not at all", "several days", "more than half the days", and "nearly every day", respectively. Higher scores mean a worse outcome.
Changes in General Anxiety Disorder-7 (GAD7) anxiety score at completion of chemotherapy assessment | Baseline assessment (prior to program) and at exercise program completion (at 24 weeks).
  General Anxiety Disorder-7 total score for the seven questions ranges from 0 (no anxiety) to 21 (highest level of anxiety). This is calculated by assigning scores of 0 (minimum), 1, 2, and 3 (maximum), to the response categories of "not at all", "several days", "more than half the days", and "nearly every day", respectively. Higher scores mean a worse outcome.
Changes in activity levels via Godin Leisure-Time Exercise Questionnaire | Baseline assessment (prior to program) and at exercise program completion (at 24 weeks).
  Godin Leisure-Time Exercise Questionnaire is used to measure a person's frequency and intensity of exercise during a typical week. A Godin Scale Score of 24 units or more is interpreted as Active, 14 - 23 units is Moderately Active, and less than 14 units is Insufficiently Active/Sedentary.
Changes in resting metabolic rate at completion of chemotherapy | Baseline and at program completion (within 4 weeks of exercise completion).
Changes in body composition at completion of chemotherapy, including fat-free mass in pounds. | Baseline and at program completion (within 4 weeks of exercise completion).
Changes in Y-Balance Test Scores at baseline and at completion of chemotherapy | Baseline and at program completion (within 4 weeks of exercise completion).
  Reach distances in three directions (anterior, posteromedial, and posterolateral) measured in centimeters.
Changes in Functional Mobility Score at baseline and at completion of chemotherapy | Baseline and at program completion (within 4 weeks of exercise completion).
  During the test, 7 movement patterns are assessed and each one is rated between 0 and 3 by an examiner. These movements include the deep squat, hurdle step, inline lunge, shoulder mobility test, active straight leg raise, trunk stability push up, and rotary stability test. A score of zero is given if any pain is felt during the movement, 1 if the subject is unable to perform the movement, 2 if the subject performs the movement through compensatory movements, and 3 if the movement is performed correctly. Each movement score is summed and a final score out of 21 is calculated. A score below 14 is felt to identify individuals at risk of injury.
Changes in phase angle at completion of chemotherapy | At program completion (at 24 weeks)
  Phase angle is calculated via bioimpedance analysis and is measured in degrees.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Champ, MD, Principal Investigator — AHN Radiation Oncology
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States